CLINICAL TRIAL: NCT06384027
Title: Acute Effects of Non-invasive Ventilation on Muscle Function Diaphragmatic and Inferior Vena Cava Distension in People Healthy
Brief Title: Effects of Non-invasive Ventilation on Function Diaphragmatic and Caval Distension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Eduardo Eriko Tenório de França, Clinical Professor, Federal University of Paraíba
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: VNI_USG_2024
Record Dates: First submitted 2024-04-17; First posted 2024-04-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Healthy
Keywords: Non-invasive ventilation; Diaphragmatic ultrasound; Inferior vena cava
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Intervention Model Description: This is a crossover, randomized study, blinded
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Spontaneous breathing (No Intervention): The volunteer will remain lying down for a period of 5 minutes in spontaneous breathing and after this period the diaphragmatic and inferior vena cava ultrasound outcomes will be evaluated.
- CPAP (Active Comparator): When using CPAP, these same outcomes will be evaluated at three different PEEP levels, namely: 5, 10 and 15 cmH2O after 5 minutes of use.
  Interventions: Other: Non-invasive ventilation
- Bilevel (Active Comparator): During the use of Bi-level, we will maintain the PEEP value at 5cmH2O and modify the pressure support (PS) ventilation values, establishing the following values: 5, 7 and 10 cmH2O of PS, with all outcomes also being evaluated at the same time. end of 5 minutes.
  Interventions: Other: Non-invasive ventilation

INTERVENTIONS:
Other: Non-invasive ventilation — Ventilation support that does not require an artificial airway that aims to reverse respiratory muscle fatigue and decrease the work of the respiratory muscles, maintaining a positive pressure, allows alveolar recruitment, preventing atelectasis and airway collapse. NIV can be administered using continuous positive airway pressure (CPAP) or two levels of airway pressure (Bi-level).
  Arms: Bilevel; CPAP

SUMMARY:
Introduction: Understanding how the applicability of non-invasive ventilation can directly affect the anatomy and diaphragmatic function, as well as the opening diameter of the inferior vena cava in healthy individuals is fundamental to knowing how this therapy can interfere with treatment results. Objective: Identify the acute effects of PEEP and ventilatory support pressure on thickening fraction, diaphragmatic mobility and vena cava distension in healthy people. Methods: This is a crossover, randomized study, blinded to the evaluator and the researcher responsible for the statistical analysis. Volunteers will undergo a NIV session, randomized into groups: CPAP, Bi-level and spontaneous breathing, without NIV support (control). The outcomes evaluated will be diaphragmatic ultrasound and inferior vena cava distensibility. The CPAP levels will be: 5, 10 and 15 cmH2O after 5 minutes of use and in the Bi-level group we will maintain the PEEP value at 5cmH2O and modify the pressure support values to the values: 5, 7 and 10 cmH2O pressure support, with all outcomes also being assessed after 5 minutes. Participants will remain in a supine position, with the right upper limb positioned behind the head, throughout the protocol and all measurements will be collected in the inspiratory and expiratory phases with volumes basal currents. For statistical analysis, intention-to-treat analysis will be employed and groups will be compared using Student's t-test, for continuous variables, or chi-square, for categorical variables. ANOVA split-plot, repeated measures for primary occurrences. Analyzes of covariance to identify differences between groups using baseline scores as covariates. Effect sizes and confidence intervals will be calculated using eta squared (η²). Expected results: Elucidate the effects of different blood pressure levels on diaphragmatic function and inferior vena cava distension.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers;
* Age equal to or over 18 years old and under 50 years old.

Exclusion Criteria:

* Cardiopathy;
* Pneumopathy;
* Participants who develop any disabling condition that prevents completion of the protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2024-04-24 (Actual); Primary Completion 2024-07-21 (Actual); Study Completion 2024-07-21 (Actual)

PRIMARY OUTCOMES:
Diaphragmatic thickening fraction | The assessment will be carried out after 5 minutes of RE, CPAP or Bilevel
  Diaphragmatic ultrasound is a useful technique for evaluating diaphragm function. To evaluate atrophy, it will be necessary to evaluate the thickening fraction (EF). A high-frequency linear transducer (7-13 MHz) will be placed over the ZA, between the eighth and ninth intercostal space, usually 0.5-2.0 cm below the costophrenic angle, between the anterior axillary line and the axillary line. medium, at a depth of 1.5 to 3 cm. The thickening fraction will be measured from the center of the pleural line to the center of the peritoneal line, at the end of expiration (Tdi-exp) and then at the end of inspiration (Tdi-insp), in modes B and M. calculated as follows:
  FE = Tdi-insp - Tdi-exp × 100 Tdi-exp

SECONDARY OUTCOMES:
Diaphragmatic mobility | The assessment will be carried out after 5 minutes of RE, CPAP or Bilevel
  Diaphragmatic mobility (MD) is measured by visualizing the hemidiaphragms through the anterior subcostal route with the convex probe below the costal margin between the midclavicular line and the anterior axillary line, the ultrasound shows the diaphragm as a deep curved structure that separates the thorax from the abdomen. To quantify mobility and diaphragmatic thickening objectively, it is necessary to evaluate at least three images and calculate the average of the MD and FE values. During the assessments, we visualize the MD during calm breathing.

OTHER OUTCOMES:
Ultrasound of inferior vena cava distension | The assessment will be carried out after 5 minutes of RE, CPAP or Bilevel
  The assessment of distension of the inferior vena cava is carried out with a convex transducer, in the subcostal window, below the xiphoid process, so that the evaluator monitors changes in diameter in real time, according to the participant's respiratory movements, thus evaluating the inspiratory and expiratory diameter of the inferior vena cava, which will later be analyzed to obtain the inferior vena cava collapsibility index:
  [(Maximum diameter - Minimum diameter) / Maximum diameter] X 100.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Paraiba, João Pessoa, Paraíba, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jansen D, Jonkman AH, Vries HJ, Wennen M, Elshof J, Hoofs MA, van den Berg M, Man AME, Keijzer C, Scheffer GJ, van der Hoeven JG, Girbes A, Tuinman PR, Marcus JT, Ottenheijm CAC, Heunks L. Positive end-expiratory pressure affects geometry and function of the human diaphragm. J Appl Physiol (1985). 2021 Oct 1;131(4):1328-1339. doi: 10.1152/japplphysiol.00184.2021. Epub 2021 Sep 2. PMID 34473571